#### הנוהל לניסויים רפואיים בבני-אדם 2020 3.1 งอเง מספר:203811 0363-20-SOR הסָכּמה מדּעת של הורי קטין להשתתפות במחקר רפואי



הטופס מנוסח בלשון זכר מטעמי נוחות בלבד אך מיועד לשני המינים.

מוצע לילדכם להצטרף לניסוי רפואי. ניסוי רפואי הוא תהליך חדשני שאינו מוכר או לא מקובל או שטרם אושר לטיפול שיגרתי בישראל ובשל כך קיימת אי ודאות לגבי בטיחותו או יעילותו. בטופס זה מוסבר על הניסוי אליו הוזמן ילדכם להצטרף. נבקשכם לקרוא את המידע בעיון ולשוחח עליו עם כל מי שתרצו: חברים, קרובי משפחה ורופאים או אנשי מקצוע בתחום הבריאות שאינם מעורבים ישירות בניסוי. מידע נוסף על הניסוי וכן מענה על שאלות ניתן לקבל מרופא הניסוי או נציגיו.

טרם ההחלטה על הצטרפות לניסוי, חשוב מאוד לדעת את הסיכונים ואת היתרונות הקיימים, כדי לקבל החלטה מושכלת. תהליך זה נקרא "הַסְכַּמֵה מִדַּעַת". כהורים אתם האחראים על מתן הסכמה בשם ועבור ילדכם.

ההסכמה להשתתפות ילדכם בניסוי נעשית מרצון החופשי וזכותכם לבחור שלא לשתף בו את ילדכם ולא לחתום על טופס ההסכמה. ניתן לפרוש מהניסוי בכל זמן, בלי לתת סיבה. להחלטתכם על סירוב או פרישה, לא תהיה השפעה שלילית על הטיפול הרפואי בילדכם כעת או בהמשך, ויוסבר לכם מהן אפשרויות הטיפול העומדות לרשותכם.

אם אתם מעוניינים לצרף את ילדכם לניסוי, תתבקשו לחתום על טופס זה. תקבלו עותק חתום לשמירה והמקור יישמר במוסד הרפואי.

ילדכם יקבל מרופא הניסוי או נציגיו, הסבר על המחקר, <u>בנוכחותכם</u>.

| שם משפחה: | :שם פרטי של הקטין |
|-----------|-------------------|
| | מס' תעודת זהות: |
| | כתובת: |
| | תאריך לידה: |

# <u>מידע על הניסוי</u> (1

הופק ע"י:ד"ר גל מאירי

0363-20-SOR מספר המחקר:

1.1) נושא הניסוי: הערכת היעילות של תוכנית התערבות מוקדמת מונחית הדרכת הורים "social ABCs" לילדים על הרצף האוטיסטי.

| תוכנית התערבות מוקדמת מונחית הדרכת הורים<br>Social ABC`s עברית | 15/12/2022 | | 4 |
|---|---|---|---|
| | Version Date תאריך גרסה | Version | גרסה |

Protocol no.0363-20-SOR



0363-20-SOR



עמוד 1 מתוך 6

5-Jun-25

| הנוהל לניסויים רפואיים בבני-אדם 2020 |
|-------------------------------------------------------|
| טופס 3.1 |
| 203811:מספר 0363-20-SOR |
| הַסְכָּמָה מִדַּעַת של הורי קטין להשתתפות במחקר רפואי |



- החוקר ד"ר גל מאירי קיבל אישור לביצוע הניסוי מוועדת הלסינקי המוסדית וממנהל המוסד הרפואי (ניסויים רפואיים בבני-אדם) המרכז הרפואי האוניברסיטאי סורוקה, בהתאם לתקנות בריאות העם (ניסויים רפואיים בבני-אדם) תשמ"א 1980.
  - 1.3) מטרת הניסוי: בדיקת יעילות התערבות מוקדמת מונחית הורים לילדים המאובחנים עם ASD
- 1.4 הטיפול בניסוי: במחקר ישתתפו ילדים שאובחנו עם אוטיזם לפני גיל 3. ההורים יונחו כיצד להעביר את ההתערבות במשך 6 שבועות. התהליך יכלול מפגשי הדרכה קבוצתיים להורים ומפגשים הדרכה פרטניים עם ההורים והילדים. ההנחיה תתבצע על ידי טניה ניצן, תמר מץ ו/או תמר דוד סטודנטיות לתואר שני ושלישי שהשלימו את תוכנית ההכשרה על ידי הוגי הגישה מהצוות הקנדי. הטיפול יועבר בתאום ותחת הנחיית הצוות של פרופ Jessica Brian 'מאוניברסיטת הולנד בלורוויו בטורונטו, קנדה. וההתערבות תתמקד ברכישת שפה ודיבור וכן ביצירת הנאה משותפת בין ההורים והילדים.
  - .1.5 מספר המשתתפים בניסוי: במחקר צפויים להשתתף 100 ילדים והוריהם.
- **1.6)** התקופה הצפויה למהלך הניסוי: במסגרת המחקר ההורים והילדים ישתתפו בתוכנית התערבות שתמשר 6 שבועות .

לפני תחילת ההתערבות, ו-12 שבועות לאחר תחילתה, הילדים יעברו הערכות שפתיות ותקשורתיות, וכן ההורים יידרשו למלא שאלונים.

1.7) שיטות הניסוי: במהלך 6 השבועות, ההורים יידרשו להשתתף בפגישה קבוצתית שבועית, וכן ב 1-2 פגישות נוספות פרטניות עם קלינאית. התוכנית הינה מובנית, וכוללת 8 יחידות, ומלווה במדריך להורים שיימסר להורים בעת תחילת ההתערבות. במפגשים הקבוצתיים הקלינאית תעביר את המידע התיאורטי, שייושם בהמשך במפגשים הפרטניים. במהלך הטיפול הקלינאית תדריך את ההורים כיצד לנהל אינטראקציות חברתיות עם ילדם בכדי להגביר את התקשורת החברתית והמילולית תוך דגש על הנאה משותפת עם ילדם.

המפגשים יתקיימו בבית החולים סורוקה, ביחידה לגיל הרך, או באופן מקוון על ידי שימוש בתוכנת ZOOM. המפגשים יוקלטו לצורך למידה וקידוד התנהגויות הילדים.

לפני תחילת תוכנית ההתערבות, ו-12 שבועות לאחר תחילת ההתערבות הילדים יעברו אבחונים סטנדרטיים, על מנת להעריך את השינויים בתחום השפה והתקשורת (אבחון שפה PLS-4 ואבחון תקשורת (אבחון שפה ADOS-2). בנוסף, ההורים יידרשו למלא שאלונים, חלקם ימולאו לפני ואחרי ההתערבות, ואחרים ימולאו רק לאחר השלמת ההתערבות.

| תוכנית התערבות מוקדמת מונחית הדרכת הורים<br>Social ABC`s | 15/12/2022 | | 4 |
|---|---|---|---|
| | Version Date תאריך גרסה | Version | גרסה |

Protocol no.0363-20-SOR





עמוד 2 מתוך 6

| הנוהל לניסויים רפואיים בבני-אדם 2020 |
|-------------------------------------------------------|
| טופס 3.1 |
| 203811:מספר 0363-20-SOR |
| הַסְכַּמֵה מִדַּעַת של הורי קטין להשתתפות במחקר רפואי |



- 1.8 מהי אחריותכם כהורים לקטין המשתתף בניסוי בהיענות לדרישות המחקר? אחריות ההורים למלא אחר כל דרישות המחקר, למלא את השאלונים לפני ואחרי ההתערבות ולהשתתף בכל המפגשים המתוכננים, כפי שיימסר בתחילת ההתערבות להורים, וכן להמשיך וליישם את ההתנהגויות הנלמדות גם מחוץ למסגרת הטיפולית. כמו כן, ההורים יידרשו להגיע עם הילד לאבחוני שפה ותקשורת לפני ואחרי ההתרבות.
- מהם הסיכונים הידועים ו/או אי הנוחות הצפויים כתוצאה מהשתתפות בניסוי? לתוכנית ההתערבות במחקר זה אין סיכונים כלשהם. אולם, ההשתתפות בתוכנית כרוכה בהשקעת זמן והתמדה כולל הקפדה על השתתפות מלאה בכל המפגשים המתוכננים. בנוסף, ההורים יידרשו לשנות את התנהגותם בבית ולהמשיך וליישם את עקרונות התוכנית במהלך השבוע בבית. כמו כל שינוי, זה ידרוש התמדה ומשמעת עצמית. בנוסף, יתכנו סיכונים שאינם ידועים/ניתנים להערכה מראש.
- 1.10) מהם היתרונות הצפויים לקטין כמשתתף או לאחרים במצבו, כתוצאה מהניסוי? תוכנית ההתערבות יכולה לתרום לשיפור ביכולות התקשורת של הילד כולל בתקשורת מילולית פונקציונלית תוך יצירת הנאה משותפת..
- האם קיימים טיפולים חלופיים? תוכנית התערבות זו הינה התערבות מונחית הורים. קיימים טיפולים אחרים שהינם התערבות ישירה מול הילד שאין מניעה לקבלם במקביל.. החוקר יסביר לכם על הסיכונים והיתרונות של אפשרויות הטיפול הזמינות עבור ילדכם.
- מהן הנסיבות בהן עלולה ההשתתפות בניסוי הרפואי להיפסק בהחלטת החוקר או היזם? ההורים יידרשו למלא שאלונים לפני ואחרי ההתערבות וכן להשתתף במספר מפגשים שבועיים ביחידה לגיל הרך בסורוקה או באמצעות התחברות במועד המפגש המתוכנן ל ."ZOOM"כמו כן, ההורים יידרשו להגיע עם הילד למפגשי ההערכה לפני ואחרי ההתערבות (אבחוני שפה ותקשורת). הורים שלא ישלימו את מילוי השאלונים ולא ישתתפו בכל המפגשים, השתתפותם במחקר תופסק.
  - מחקר זה אינו כולל איסוף רקמות / דגימות (2

# <u>מידע כללי</u> (3

הופק ע"י:ד"ר גל מאירי

- 08- בכל בעיה הקשורה לניסוי הרפואי תוכלו לפנות לחוקר, בכל שעות היממה בטלפון שמספרו: -08 (3.1 בכל מקרה של בעיה רפואית, פציעה או אירוע בריאותי אחר בתקופת הניסוי עליכם 6244306 בכל מקרה של בעיה רפואי מתאים וכן פרטים נוספים על זכויותיכם בהקשר זה.
- החוקר יעביר מידע על השתתפות ילדכם במחקר לרופא המטפל שלו בקהילה לצורך ידיעה ומעקב (3.2 רפואי. אם במהלך הניסוי יתגלו ממצאים רפואיים בעלי משמעות קלינית, שלא היה ידוע עליהם קודם,

| תוכנית התערבות מוקדמת מונחית הדרכת הורים<br>Social ABC`s עברית | 15/12/2022 | | 4 |
|---|---|---|---|
| | Version Date תאריך גרסה | Version | גרסה |

עמוד 3 מתוך 6

Protocol no.0363-20-SOR

Matarot Helsinki



5-Jun-25

אנא חשוב על הסביבה לפני הדפסת המסמר

0363-20-SOR

| הנוהל לניסויים רפואיים בבני-אדם 2020 | |
|-------------------------------------------------------|-------------|
| 3.1 งมเช | |
| מספר:203811 | 0363-20-SOR |
| הַסְכָּמָה מְדַּעַת של הורי קטין להשתתפות במחקר רפואי | |



המידע יימסר לרופא בקהילה. תוצאות חיוביות על מחלות החייבות בדיווח על פי חוק יישלחו למשרד הבריאות (לדוגמה: צהבת, שחפת, חצבת, HIV וכד').

- 3.3) מידע חדש, שיכול להשפיע על ההחלטה להשתתף או להמשיך בניסוי, יועבר לידיעתכם בהקדם.
- במסגרת המחקר, יתכן ותתבקשו לענות על שאלון. אתם יכולים לבחור לא לענות על כל השאלות (3.4 בשאלון או על חלק מהן אך קחו בחשבון כי השתתפותכם במחקר תופסק.
- יזם הניסוי פרופ' אילן דינשטיין משלם למוסד הרפואי את העלויות הכרוכות בביצוע הניסוי. לחוקר יש זיקה ליזם הניסוי, פרופ. אילן דינשטיין אחד מחוקרי המשנה הוא יזם הניסוי.
  - . יזם הניסוי והמוסד הרפואי דאגו לכיסוי ביטוחי במקרה של נזק הנגרם מביצוע הניסוי.
- יתכן והמחקר ירשם באתר המחקרים הקליניים של משרד הבריאות: MyTrials. האתר לא יכלול מידע שיכול לזהות את ילדכם. תוכלו לערוך חיפוש באתר זה בכל עת.

#### שמירה על פרטיות וסודיות המידע (4

- במחקר אליו התבקשתם לצרף את ילדכם נאסף מידע רפואי ואישי כחלק מהניסוי. מידע זה נשמר ברשומה רפואית ובאחריות הצוות המטפל בילדכם לשמור על סודיות רפואית. זכותכם לקבל מידע מהרשומה הרפואית בהתאם לחוק זכויות החולה. אם ידוע לכם שהמידע ברשומה הרפואית שגוי או חלקי עליכם ליידע את הצוות המטפל בילדכם.
- 4.2) ברשומה הרפואית ישמר מידע כגון: תוצאות בדיקות רפואיות, מתן תכשירים, אביזרים או משתלים, ביצוע טיפולים או פרוצדורות ניסיוניות וכדומה.
- הסכמתכם לצרף את ילדכם לניסוי הינה הסכמה גם לכך שמידע רפואי ואישי הנאסף במהלך הניסוי יועבר לגורם חיצוני, שיעשה בו שימוש לעיבוד הנתונים. המידע יועבר לגורם החיצוני רק כשהוא מקודד. המידע לא יכלול: שם, שם משפחה, מספר תעודת הזהות, כתובת המגורים או מספר מזהה אחר שניתן לילדכם על ידי רשויות המדינה.
- ככלל, מידע מקודד נחשב מידע הניתן לזיהוי. הקשר בין הקוד והפרטים המזהים של ילדכם ישמר אצל החוקר הראשי בארץ בצורה מאובטחת. במקרים מסוימים תתאפשר פתיחת הקוד על ידי החוקר.
- 4.4) הנתונים והמידע המקודדים הללו יישמרו על ידי היזם לפרק זמן המוגדר בחוק (לפחות 15 שנה מתום המחקר).
- (למשל: למשל: אות צפייה, לצורכי אימות שיטות הניסוי הרפואי והנתונים, יינתנו לגורמים מורשים בלבד (למשל: נציגים מוסמכים של היזם, ועדת הלסינקי, הגוף המבקר במוסד הרפואי ופקחים של רשויות בריאות). גישה זו למידע הרפואי תבוצע, באמצעות החוקר, ובהתאם לחוקים ולנהלים של שמירת סודיות.
  - . פרטים מזהים של ילדכם לא יופיעו באף פרסום מדעי או אחר (4.6

| תוכנית התערבות מוקדמת מונחית הדרכת הורים<br>Social ABC`s עברית | 15/12/2022 | | 4 |
|---|---|---|---|
| | Version Date תאריך גרסה | Version | גרסה |

Protocol no.0363-20-SOR

Matarot Helsinki



0363-20-SOR



עמוד 4 מתוך 6

5-Jun-25

הופק ע"י:ד"ר גל מאירי

# הנוהל לניסויים רפואיים בבני-אדם 2020 טופס 3.1 מספר:0363-20-SOR הַסְכָּמָה מָדַעָת של הורי קטין להשתתפות במחקר רפואי



### פרישה מהניסוי הרפואי (5

בכל שלב של הניסוי זכותכם להחליט על פרישה ממנו על ידי הודעה לחוקר הראשי או נציגו. אתם לא חייבים להסביר מדוע פרשתם. החוקר רשאי לעשות שימוש רק בדגימות ו/או בנתונים מקודדים שנאספו עד למועד הפרישה.

מהרגע שהודעתם על פרישה מהניסוי לא ייאסף על ילדכם מידע נוסף. יחד עם זאת, אם יתקבל מידע בעל משמעות רפואית לגבי ילדכם או לגבי בני משפחתכם ייצרו איתכם קשר. זכותכם לסרב לקבל את המידע.

## [מידע על פוריות, פריון בעתידי / הריון / עובר או תינוק יונק:] (6

לא רלוונטי

# :<u>תיעוד הסכמה</u> (7

שני הורי הקטין הם האחראים על מתן הסכמה בשמו ועבורו ברוח חוק הכשרות המשפטית והאפוטרופסות, תשכ"ב-1962.

<u>הורי המשתתף</u>: בחתימתי אני מצהיר כי קראתי את התוכן של מסמך זה, הוסבר לי על הניסוי ואני מסכים שילדי ישתתף בו.

| <b>שם ההורה</b> (פרטי ומשפחה): | חתימה: | תאריך ושעה: |
|--------------------------------|--------|-------------|
| שם ההורה (פרטי ומשפחה): | חתימה: | תאריך ושעה: |

#### משתתף שמלאו לו 16 שנים (כאשר יש בדיקות גנטיות):

קיבלתי הסבר על הניסוי ואני מסכים להשתתף בו.

| תוכנית התערבות מוקדמת מונחית הדרכת הורים<br>Social ABC`s עברית | 15/12/2022 | | 4 |
|---|---|---|---|
| | Version Date תאריך גרסה | Version | גרסה |

Protocol no.0363-20-SOR





עמוד 5 מתוך 6

# הנוהל לניסויים רפואיים בבני-אדם 2020 טופס 3.1 מספר:203811 מָסָכֶּמָה מִדַּעַת של הורי קטין להשתתפות במחקר רפואי

| www.health.gov.il | | |
|---|---|---|
| | המינהל לטכנולוגיות רפואיות ותשתיות<br>אגף הרוקחות <mark>המחלקה לניסויים קליניים</mark><br>Clinical Trials Department | משרד<br>הבריאות<br>לחיים בריאים יותר |

חתימה: תאריך ושעה:

<u>החוקר המסביר</u>: בחתימתי אני מצהיר כי הסברתי להורי הקטין בעל פה על הניסוי בהתאם לכתוב בטופס זה. אני סבור שההורים הבינו את הנאמר, היה להם מספיק זמן לקרוא את הטופס והם הביעו את הסכמתם לצרף את ילדם לניסוי.

בנוסף, אני מצהיר כי הסברתי למשתתף הקטין בנוכחות הוריו על הניסוי והוא הביע את רצונו להשתתף בניסוי.

| | חתימה: | שם (פרטי ומשפחה): |
|--------------------------|--------|---------------------------------------|
| (כולל חותמת ומספר רשיון) | ) | · |

<u>עד בלתי תלוי</u>\*: אני החתום מטה, נכחתי במשך ההסבר על הניסוי הרפואי, מאשר כי התוכן של מסמך זה נמסר בעל-פה בנוכחותי להורים ולילדם, התרשמתי שהם הבינו את ההסבר ושמעתי שהם הביעו הסכמתם בעל-פה לצרף את ילדם לניסוי.

| חתימה:תאריך ושעה: | שם (פרטי ומשפחה): |
|-------------------|-------------------|
|-------------------|-------------------|

| תוכנית התערבות מוקדמת מונחית הדרכת הורים<br>Social ABC`s עברית | 15/12/2022 | | 4 |
|---|---|---|---|
| | Version Date תאריך גרסה | Version | גרסה |

Protocol no.0363-20-SOR



שם הילד (פרטי ומשפחה):

0363-20-SOR

5-Jun-25

לשימוש רק במקרה שההורים אינם מסוגלים לקרוא את טופס ההסכמה מדעת (לוקים בראייתם או אינם יודעים קרוא וכתוב) או במצב של דחיפות רפואית (לפי הגדרת החוק). העד הבלתי תלוי חייב להיות נוכח במשך ההסבר על הניסוי הרפואי.